CLINICAL TRIAL: NCT01521598
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo Controlled Study Assessing the Efficacy and Tolerability of SKL11197 for the Pain of Diabetic Peripheral Neuropathy
Brief Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo Controlled Study for the Pain of Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SKL11197C006
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-05

CONDITIONS: Painful Diabetic Neuropathy
Keywords: Diabetic Peripheral Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SKL11197 (Experimental): This arm is the experimental drug (SKL11197) arm. Patients will be randomized to this arm.
  Interventions: Drug: SKL11197
- Placebo (Placebo Comparator): This arm is the placebo comparator arm. Patients will be randomized to this arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SKL11197 — SKL11197 drug product contains 150 mg of active ingredient. Dosing will be three times per day.
  Arms: SKL11197
Drug: Placebo — This is the placebo. Patients will be randomized the placebo.
  Arms: Placebo

SUMMARY:
Primary Objective: To evaluate the efficacy of SKL11197 for the treatment of diabetic peripheral neuropathy pain (DPN).

Secondary Objective: To evaluate the safety and tolerability of SKL11197 in subjects with painful diabetic peripheral neuropathy.

Primary Efficacy Endpoint: The primary efficacy outcome variable will be the time to exit from the double-blind phase because of inadequate pain relief.

DETAILED DESCRIPTION:
This study is a double-blind, placebo controlled study with three phases;

1. a pre-study medication washout/screening phase upto 3 weeks
2. a 3-week, open label phase
3. a 6-week double-blind phase At the end of 3-week in the open label phase, subjects may enter the double-blind phase if they meet the eligibility criteria.

Eligible subjects will be randomized in a blinded fashion either to continue with SKL11197 at 300 mg TID or to take the same number of placebo capsules.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Diagnosis of Type 1 or Type 2 diabetes mellitus for at least 1 year
3. At least moderate pain, ≥ 40mm on a 100mm VAS at the end of washout phase (in absence of any analgesic);
4. HbA1c < 12 % at Screening
5. Daily pain attributed to diabetic neuropathy for least 3 months prior to Screening on the basis of history and physical examination documenting peripheral neuropathy.
6. Pain from diabetic neuropathy should be identifiable by the subject. Pain must involve the lower extremities and be bilateral.
7. Females must be of non-childbearing potential (defined as either surgically sterile or at least one year postmenopausal, Menopause is defined as 1 year since last menstrual period with associated subjective sensations), or,
8. If capable of bearing children, females must use a double-barrier method of contraception, or an intrauterine device. Females capable of bearing children must have negative serum pregnancy (beta-HCG) test at Screening and negative urine pregnancy on Day 1.

Exclusion Criteria:

1. Pregnant or lactating females
2. Subjects with BMI over 40
3. Pain due to symptomatic peripheral vascular disease (e.g. intermittent claudication)
4. Subjects with known clinically significant decreased blood flow to the extremities
5. Subjects cannot have pain from other sources that can confuse the assessment of the diabetic neuropathic pain
6. Peripheral neuropathy attributable to other causes such as alcoholism, connective tissue disease, or toxic exposure;
7. Have profound autonomic dysfunction, or brittle diabetes;
8. Evidence of amputations (including toes), open ulcers, or Charcot joint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Relief of diabetic neuropathy pain | 24 hours

SECONDARY OUTCOMES:
Average daily pain score | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kamin, M.D., Study Director — SKLSI (Sponsor)
Locations (13):
- United States (13):
  - Neurology Clinic, P.C., Northport, Alabama
  - Principals Research Group, Hot Springs, Arkansas
  - Clinical Trials, Inc., Little Rock, Arkansas
  - Collaborative Neuroscience Network, Inc., Long Beach, California
  - Neurological Research Institute, Santa Monica, California
  - Renstar Medical Research, Ocala, Florida
  - Comprehensive Clinical Development, St. Petersburg, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - International Clinical Research Institute, Leawood, Kansas
  - Michigan Head Pain & Neurological Institute., Ann Arbor, Michigan
  - Creighton Diabetes Center, Omaha, Nebraska
  - Sunstone Medical Research, LLC, Medford, Oregon
  - Nerve and Muscle Center of Texas, Houston, Texas